CLINICAL TRIAL: NCT04554199
Title: Evaluation of Changes in Brain Activity and Cognitive Function of Diabetic Patients Wearing Removable Partial Dentures
Brief Title: Brain and Cognitive Function of Patients With RPD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Research Centre, Egypt (Other)
Responsible Party: Principal Investigator, Asmaa Nabil Elboraey, Associate Professor, National Research Centre, Egypt
Allocation: Non-Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 16-086
Record Dates: First submitted 2020-08-29; First posted 2020-09-18 (Actual); Last update posted 2020-09-18 (Actual); Status verified 2020-09

CONDITIONS: Missing Posterior Occlusal Contact
Keywords: Removable partial dentures; Electro-encephalogram; Mini mental state examination; Controlled type 2 diabetes.

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Participants, as well as the investigating dentist are blind to the result obtained from the EEG recording. The statistician is also unaware of the EEG .
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EEG and MMSE measurements before receiving RPD (Experimental): EEG and MMSE were measured for all participant before wearing the removable partial dentures.
  Interventions: Device: Flexible partial denture
- EEG and MMSE measurements after receiving RPD (Experimental): EEG and MMSE were measured for all participant after wearing the removable partial dentures
  Interventions: Device: Flexible partial denture

INTERVENTIONS:
Device: Flexible partial denture — removable partial dentures (RPDs) were fabricated using thermoplastic resins (flexible RPDs). EEG and MMSE were evaluated before denture delivery and after one month of denture wear.

SUMMARY:
To evaluate the influence of restoring lost posterior occlusal contacts with removable partial denture (RPD) on the brain activity and cognitive function in controlled type 2 diabetic patients

ELIGIBILITY:
Inclusion Criteria:

* Loss of posterior occlusal contact unilaterally or bilaterally in both maxilla and mandible.
* No previous partial dentures experience.
* Nonsmokers.
* Skeletally Angle's class I.
* Controlled type 2 diabetes.

Exclusion Criteria:

* History of brain diseases (e.g. cerebral infarction, and Alzheimer's).
* Neuromuscular disorders.
* Temporomandibular joint disorder.
* Psychiatric illness.
* Participants with parafunctional oral habits.

Ages: 40 Years to 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Males sex were selected to avoid the possible influence of hormonal imbalance in female on brain activity and cognitive function.
Enrollment: 30 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2019-05-01 (Actual); Study Completion 2019-07-01 (Actual)

PRIMARY OUTCOMES:
Brain activity measurement in controlled type 2 diabetic patients wearing RPD. | For each participant the RPD should be worn for one month.
  RPDs were fabricated for each participant using thermoplastic resin. The brain activity was assessed using EEG by measuring the alpha waves (Dα/Hz) in controlled type 2 diabetic patients wearing RPDs. EEG records were obtained before denture delivery and one month after denture wear.
Cognitive function assessment in controlled type 2 diabetic patients wearing RPD. | For each participant the RPD should be worn for one month.
  For the same participates the cognitive function was assessed via MMSE questionnaire. MMSE consists of 12 questions with maximum scoring of 30. The measurements were obtained before denture delivery and one month after denture wear.

CONTACTS AND LOCATIONS:
Locations (1):
- National Research Centre, Cairo, Dokki, Egypt

IPD SHARING:
Plan to Share IPD: No